CLINICAL TRIAL: NCT04865939
Title: A Randomized Trial Comparing Intravesical Gemcitabine to Continuous Bladder Irrigation With Sterile Water to Prevent Bladder Cancer Implantation in Patients Undergoing Excision of Upper Tract Urothelial Carcinoma
Brief Title: Gemcitabine Versus Water Irrigation in Upper Tract Urothelial Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, yair lotan, Professor and Chief of Urologic Oncology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2021-0402
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Cancer of Renal Pelvis; Urothelial Carcinoma Ureter
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: randomized, single-blinded controlled noninferiority trial
Who Masked: Participant
Masking Description: Participants will not be informed of group allocation. Blinding treating clinicians is impractical due to the techniques used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- gemcitabine (Active Comparator): intravesical instillation of gemcitabine (1 g in 50 mL saline) with dwell time of 1 - 3 hours
  Interventions: Drug: Gemcitabine
- sterile water irrigation (Experimental): intravesical continuous bladder irrigation with sterile water for 1 - 3 hours and a total instilled volume of approximately 4 - 16 liters
  Interventions: Procedure: sterile water irrigation

INTERVENTIONS:
Procedure: sterile water irrigation — Continuous irrigation of bladder with sterile water during surgery (prior to entry into bladder).
  Arms: sterile water irrigation
Drug: Gemcitabine — Intravesical gemcitabine instilled into bladder during surgery (drained prior to entry into bladder).
  Arms: gemcitabine

SUMMARY:
There is a high rate of intravesical (bladder) recurrence following extirpative surgery for upper tract urothelial carcinoma. There is no single established standard of care for prevention of intravesical recurrence; however, one protocol in common use involves the use of intravesical gemcitabine instilled into the bladder during surgery and prior to entry into the bladder. There are barriers to the use of gemcitabine, especially at lower volume centers. Some evidence suggests that intravesical irrigation with sterile water has equivalent efficacy to intravesical chemotherapy in prevention of recurrent bladder cancer following transurethral resection of bladder tumors (TURBT). This study is intended to compare recurrence rates using intravesical gemcitabine (as a pseudo-standard of care) and continuous bladder irrigation with sterile water.

DETAILED DESCRIPTION:
Upper tract urothelial carcinoma is a relatively rare disease, accounting for 5-10% of urothelial malignancies. Following radical nephroureterectomy (RNU), recurrence of urothelial carcinoma in the bladder (UCB) is reported in up to 50% of cases. Although the mechanism of bladder cancer recurrence following RNU is still controversial, recent evidence suggest that these tumors have similar clonal origin to upper tract tumors, supporting the theory of downstream seeding; specifically, that manipulation of the upper tract during surgery results in shedding of tumor cells which then implant in the bladder and give rise to bladder tumors.

Different strategies have been suggested to reduce UCB recurrence rates following RNU. Early clipping of the ureter distal to the tumor may prevent seeding and reduce UCB recurrence, while the correct technique for bladder cuff resection remains debatable. A single, post-operative, prophylactic intravesical chemotherapy instillation (pIVC) has been shown to reduce recurrence rates following resection of UCB. Specifically, two prospective studies have evaluated the use of pIVC using mitomycin-C (MMC) or pirarubicin (THP) following RNU, showing a 11-25% absolute reduction in the risk of UCB recurrence. The safety of pIVC has previously been reported by Moriarty et al. with no directly associated adverse events. The investigators' group also compared bladder recurrence rates in patients who received intraoperative or postoperative pIVC. In this cohort, 12- and 24-month recurrence rates in the I-pIVC groups were 10.8% and 14.4%, respectively, with a favorable safety profile. Current practice at this institution, which is widely employed at many centers but is not supported by Level I evidence, is to instill gemcitabine into the bladder intraoperatively and to allow it to dwell within the bladder until excision of the ureter, at which time the gemcitabine is drained prior to entry into the bladder.

Despite its demonstrated benefits, there appears to be considerable underutilization of pIVC for various reasons. Based on a national survey in the United States, less than 50% of urologic oncologists use pIVC, mainly due to concerns including lack of evidence, fear of extravasation and office infrastructure. While educational measures should be taken to increase urologists' awareness of the importance and high level evidence supporting the use of pIVC, other concerns, such as extravasation and logistical issues (which may include office infrastructure, availability of chemotherapeutic agents outside of a hospital setting, availability of trained personnel, etc.).

A possible alternative to pIVC that would circumvent logistical, availability-, and toxicity-based concerns is the use of intravesical continuous bladder irrigation (CBI) with sterile water. In this method, a multi-way urinary catheter is placed in the bladder which allows water to be irrigated into the bladder while simultaneously and freely draining out via a separate lumen, allowing the bladder to be continuously irrigated with sterile fluid. In this setting, irrigation would be initiated at the start of the surgical procedure and would be terminated and the bladder drained immediately prior to entry into the bladder at the time of excision of the distal ureter. There have been several studies that have demonstrated the ability of hypotonic fluid (e.g., sterile water) to kill bladder tumor cells. Distilled water irrigation has shown to delay tumor recurrence of bladder cancer by osmolysis of tumor cells. A prospective, randomized, open-label, two-arm, single-center, pilot study compared continuous sterile water irrigation to a single dose intravesical of mitomycin C after transurethral resection of bladder tumors (TURBT) and found recurrence-free rates for MMC and continuous sterile water irrigation groups were 47.1% and 52.6%, respectively. Another study investigated the results of bladder irrigation with water for injection after TURBT. A total of 239 patients (158 with single tumors, group A, and 81 with multiple tumors, group B) received continuous intravesical postoperative irrigation with water. Recurrence-free rate for those patients who received only intravesical irrigation with water was 75.8%, 66.2% and 63.2% at the 1st, 2nd and 3rd year of follow up, respectively. A systemic review of the literature evaluated bladder irrigation after TURBT. There were 6 studies, including 1515 patients of which 361 had saline irrigation and 463 had sterile water. There was no significant difference between IVT chemotherapy, saline and sterile water groups regarding to the median RFS at 1 year [IVT: 81%, IQR (77.70, -81.00), sterile water: 74%, IQR (63.3-74.9), saline: 76.7% IQR (76.0, 77.7), p = 0.21]. Adverse events were more frequent amongst patients in the IVT chemotherapy group in comparison to the saline or water groups.

In this study, it is hypothesized that intraoperative continuous bladder irrigation with sterile water is noninferior to intravesical instillation of gemcitabine. If the two regimens are substantially equivalent, irrigation with water would be considered a superior option due to greater simplicity, wider availability, and reduced risk of toxic exposure to the patient and operating room staff.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven UTUC with plan for excisional surgery (distal ureterectomy or nephroureterectomy) with curative intent
* Age 18 - 90 years
* Life expectancy > 1 year
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Concurrent or prior diagnosis of bladder cancer with a disease-free interval of less than three years.
* Synchronous bilateral upper tract urothelial carcinoma (prior history of contralateral UTUC is permissible with a disease-free interval of more than three years).
* Plan for radical cystectomy.
* Small bladder capacity (< 100 mL).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or other agents used in study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
intravesical recurrence | 1 year
  rate of biopsy proven intravesical recurrence of urothelial carcinoma
intravesical recurrence | 2 years
  rate of biopsy proven intravesical recurrence of urothelial carcinoma

SECONDARY OUTCOMES:
treatment-related associated adverse event rate | 30 days
  rate of CTCAE grade 1-3 complications

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freifeld Y, Ghandour R, Singla N, Woldu S, Bagrodia A, Lotan Y, Rapoport LM, Gazimiev M, Delafuente K, Kulangara R, Robyak H, Petros FG, Raman JD, Matin SF, Margulis V. Intraoperative prophylactic intravesical chemotherapy to reduce bladder recurrence following radical nephroureterectomy. Urol Oncol. 2020 Sep;38(9):737.e11-737.e16. doi: 10.1016/j.urolonc.2020.05.002. Epub 2020 Jul 5. PMID 32641241